CLINICAL TRIAL: NCT02111733
Title: Is High Sensibility Troponins a Dialysable Marker in Hemodialysis Patients and Does it Have Prognostic Value?
Acronym: TnT-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TnT-HD
Record Dates: First submitted 2013-12-10; First posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hs-TnT (Experimental): Hs-TNT dosage
  Interventions: Other: Hs-TNT dosage

INTERVENTIONS:
Other: Hs-TNT dosage — Bloodwork before and after hemodialysis for high sensibility troponins T blood level

SUMMARY:
Evaluation of High sensibility troponin levels modification by hemodialysis in terminal renal failure patient at Sherbrooke University Hospital Center as determined by serial measurements. Verification of potential effects of these levels and their variation as predictors of cardiovascular outcomes and events at 6 and 12 months.

DETAILED DESCRIPTION:
Recruiting of hemodialysis patients of the nephrology renal supplementation clinics at Sherbrooke University Hospital Center to measure three blood level of high-sensibility troponins before and after standard dialysis. Verification on the variation of these levels after dialysis. Follow-up at 6 and 12 months of the patient for Cardiovascular events and death and verification of a possible predictive value of troponin blood levels for these events.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years, no symptoms, over 1 months of hemodialysis

Exclusion Criteria:

* 1 or more in the last month; Acute coronary syndrome, Heart failure decompensated, Myo or Pericarditis, Pulmonary embolism, Sepsis/shock, Stroke or transient ischemic attack, Malignant high blood pressure, Arrythmia, electrical cardio-version, major trauma, significant burnings (>25%), Chemotherapy, Cardiovascular surgery, percutaneous angio-intervention,
* Chronic systemic disease (sarcoidosis, amyloidosis, LED, Etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
High sensibility troponins T blood level variation | 1 week
  Verification of high sensibility troponins T blood after classical hemodialysis compared to pre-treatment levels.

SECONDARY OUTCOMES:
Prognostic value of high sensibility troponins T blood level variation | at 6 and 12 months
  Evaluation of a potential prognosis value of high sensibility troponins T blood levels and its variation after hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Nguyen, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (2):
- Canada (2):
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec